CLINICAL TRIAL: NCT07397273
Title: Effects of Alpha-GPC on Lower Body Muscular Performance and Activation.
Brief Title: Acute Effects of Alpha-glycerylphosphorylcholine (A-GPC) on Lower Body Muscular Performance.
Acronym: A-GPC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Clayton Camic, Professor, Northern Illinois University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #HS25-0236
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult Participants
Keywords: supplementation; isometric; electromyography; Wingate Anaerobic Test; muscular power; ergogenic aid
MeSH Terms: interventions — Glycerylphosphorylcholine; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, within-subjects, crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement group (Experimental): Oral Alpha-GPC (900 mg)
  Interventions: Dietary Supplement: L-Alpha glycerylphosphorylcholine
- Placebo group (Placebo Comparator): Oral microcrystalline cellulose
  Interventions: Dietary Supplement: Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: L-Alpha glycerylphosphorylcholine — Oral, 900 mg, single dose study
  Arms: Supplement group
Dietary Supplement: Microcrystalline Cellulose — Oral, 900 mg, single dose study
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
The purpose of the present study was to examine the effectiveness of acute A-GPC supplementation on upper and lower body muscular strength, endurance, power, and global levels of activation.

DETAILED DESCRIPTION:
Nutritional supplementation has become an integral component of training and competition strategies for athletes attempting to maximize their exercise performance capabilities. Multi-ingredient pre-workout supplements are commonly utilized products included in this process and designed to be ingested prior to training or sport for the purpose of enhancing factors such as muscular strength and endurance, aerobic capacity, and feelings of energy, alertness, and focus (Jagim et al., 2019). Although the ergogenic effects of various pre-workout supplements have recently been examined in numerous studies (Harty et al., 2022), comparing the results among these products remains challenging due to different ingredients formulations, dosages, proprietary blends, and inclusion of a large number of ingredients (Jagim et al. 2019) that have not been assessed for their isolated effectiveness (Harty et al., 2022).

Alpha-glycerlphosphocholine (A-GPC) is one of those ingredients found in numerous pre-workout supplements and energy drinks with limited data on its individual ergogenic effects. Specifically, A-GPC (also known as alpha-GPC and choline alfoscerate) is a semi-synthetic derivative of lecithin and an esterified form of choline (Brownawell et al. 2011) that is considered one of the most used variants due to its high choline content and its ability to cross the blood-brain barrier (Kansakar et al., 2023). When orally administered, A-GPC is converted to phosphatidylcholine, an active form of choline that yields an A-GPC to choline ratio of 1.0/0.4 mg (Abbiati et al. 1993; Bellar et al. 2015; Brownawell et al. 2011; Govoni et al. 1992; Traini et al. 2013). Choline is a critical component of the neuronal phospholipid bilayer and an important nutrient for the human body involved in the function of numerous organs like the liver, kidney, spleen, and lungs (Kansakar et al., 2023; Abbiati et al., 1993; Traini et al., 2013; Govoni et al., 1992). Moreover, choline is a precursor to acetylcholine (ACh), a diverse neurotransmitter in areas including the hippocampus, cerebral cortex, and neuromuscular junction where it functions in a crucial role for memory formation, cognitive function, and muscle activation through the transfer of action potentials between neurons and muscle fibers (Kansakar et al. 2023). Based on the latter mechanism, it has been suggested (Bellar at al., 2015; Markus et al. 2017; Zeigenfuss et al., 2008) that increased ACh formation from A-GPC supplementation may result in an augmented signal for contraction, thereby leading to greater muscular strength and power during intense exercise. In addition, increased use of A-GPC in animal models has shown the potential of enhanced effects on cognitive function, likely due to the increased cholinergic transmission, dopaminergic neurotransmission, and the serotonergic system, which are closely linked to increased motivation and decreased anxiety (Tayebati et al., 2013; Salamone et al., 1994; Robinson et al., 2005; Bromberg-Martin et al., 2010). Based on these potential mechanisms, acute supplementation of A-GPC may have potential for augmenting high-intensity performance.

The majority of previous studies on A-GPC supplementation have examined its effect on cognitive functions and physical performance. Recent findings reported increased self-reported motivation, yet no difference in depression, anxiety, and mood with the ingestion of 400 mg A-GPC (Tamura et al., 2021). In addition, A-GPC supplementation has been found to improve reaction time for psychomotor vigilance, Stroop, and serial-subtraction tests at dosages ranging from 200- 630 mg (Marcus et al., 2017; Kerksick, 2024; Parker et al., 2016), whereas, at dosages of 500 mg resulted in no difference of reaction time, visual and verbal memory during an ImPACT test (Bunn et al., 2018). While prolonged supplementation of A-GPC has been shown to improve peak force in isometric contractions (Bellar et al., 2015), acute supplementation of A-GPC has demonstrated conflicting results for its ergogenic effects during physical activity. Previous findings have reported benefits of A-GPC supplementation to increase isometric strength and peak force with a 600 mg dosage (Ziegenfuss et al., 2008; Barzanjeh et al., 2022); however, other studies found contrasting evidence reporting no effect in power, average force, and work capacity with similar dosages (315-630mg) (Bunn et al., 2018; Kerksick, 2024). It is possible findings of A-GPC have been inconsistent, due to the wide range of dosages administered in each study ranging from 200 mg to 1g and their differences in concentration (50-99%), its combination with other substances, and protocol of exercise (Parker et al., 2016; Barzanjeh et al., 2022). Examples of these noted reasons can be observed in many studies that used the protocol of 60 minutes of ingesting the supplement prior to exercise testing, following the response in growth hormone (GH) release found by Ceda et al., (1991) where when 1 g of A-GPC was intramuscularly injected the peak GH release was 60 min after injection. This, however, was a different method of ingesting the supplement than most individuals have access to. Ziegenfuss et al., (2008), reported the GH response to oral ingestion of 600 mg A-GPC had a peak GH release after 90 minutes post-consumption. With the increased popularity of A-GPC being used in acute supplementation, more research is needed to ensure a proper dosage, impact on exercise performance, and its effect on muscle activation (Marcus et al., 2017). Due to these reasons, the purpose of the present study was to examine the effectiveness of acute A-GPC supplementation on upper and lower body muscular strength, endurance, power, and global levels of activation.

Previous studies of A-GPC have examined the effects of psychomotor vigilance and its role in improving cognitive functions (i.e. mood, motivation, memory, alertness, reaction time) (Marcus et al., 2017, Tamura et al., 2021, Kerksick, 2024). In a study by Tamura et al. (2021), it was discovered that after a dosage of 400mg of A-GPC for two weeks, self-reported motivation improved, potentially due to the increased cholinergic transmission. Other evidence has been reported that in two different acute doses of A-GPC (250 mg and 500 mg) free serum choline levels increased, also resulting in improved reaction time (Marcus et al., 2017). Other studies have discovered evidence of A-GPC resulting in no significant differences when compared to the placebo or other supplements. The first study by Bunn et al., (2017), delved into an acute dose of 500 mg of A-GPC and its combination with 250 mg of uridine-5'-monophosphate, and 1500 mg DHA, finding no difference in verbal memory, visual memory, visual motor speed, and reaction time. Another study examined 20 healthy individuals in a serial subtraction test resulting in improved times by 18.1% and 10.5% compared to caffeine and placebo groups, respectively. (Parker et al., 2016). On the other hand, in terms of physical performance, choline supplementation has been proven to be effective after prolonged use. In a study conducted by Lee et al., (2023), 37 50-69 year old participants followed a 12-week resistance training protocol where participants were split into three groups all taking different dosages of choline (low, medium, high), resulting in a significant change in composition strength for the medium and high groups compared to the low. Comparatively, it has been shown that after chronic use of 600 mg A-GPC supplementation, there was a significant increase in peak force from baseline compared to the placebo group in an isometric mid-thigh pull; though in the same study, it was shown that after an acute dosage of the choline-rich supplement showed no significant measures in isometric strength for the upper body (Bellar et al., 2015). More evidence on ergogenic effects of 600 mg A-GPC has been found through the investigation by Ziegenfuss et al., (2008), where 7 resistance-trained men improved peak bench press force by 14% when compared to the placebo group. Another study investigating a higher dosage of A-GPC (1000 mg) has been found to increase peak power, mean power, and fatigue index whilst lowering systolic blood pressure, diastolic blood pressure, and heart rate in recovery with overweight and obese women after different frequency sprint interval exercise (Barzanjeh et al., 2022). These studies contribute to the suggestion of acute dosages be over 500 mg, because in the study by Bunn et al., (2017), there was no significant difference in power output or work capacity through the means of vertical jump and bench press. Though it has been seen in a multiple-ingredient supplementation study consisting of l-citrulline, branched chain amino acids, and 300 mg of A-GPC, provided a significantly higher peak power output of 11% in a 20-km timed trial on a cycle ergometer by 30 male trained cyclists, but this could be due to the known ergogenic effects of l-citrulline and its role in nitric oxide production (Harrington et al., 2017).

Through the popularity of A-GPC being used in acute supplementation, more research is needed to ensure a proper dosage and its impact on exercise performance. Many studies used the protocol of 60 minutes of ingesting the supplement prior to exercise testing, following the response in growth hormone (GH) release found by Ceda et al., (1991) where when 1 g of A-GPC was intramuscularly injected the peak GH release was 60 min after injection. This, however, was a different method of ingesting the supplement than most individuals have access to. Ziegenfuss et al., (2008), reported the GH response to oral ingestion of 600 mg A-GPC had a GH release after 90 minutes post-consumption. Since prior research has looked at numerous dosages and different means of exercise, the purpose of this study was to evaluate the efficacy of A-GPC shown in anaerobic power, strength, and endurance through electromyography (EMG) in healthy, resistance trained men.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally-trained males, college-aged

Exclusion Criteria:

* If the subjects report: 1) cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders; 2) use of any medications; 3) use of nutritional supplements; 4) habitual use of caffeine (≥1 caffeinated beverage per day); 5) participation in another clinical trial or investigation of another nutritional product within 30 days of screening/enrollment.

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction | Approximately 90 minutes post-ingestion of condition
  MVIC of leg extensors at 120 degrees between thigh and leg
Muscle Activation | Approximately 90 minutes post ingestion
  EMG amplitude during MVIC

SECONDARY OUTCOMES:
Wingate Anaerobic Test | Approximately 100 minutes post-ingestion of condition
  Peak, mean, minimum power and fatigue index

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Camic, PHD, Principal Investigator — Northern Illinois University
Locations (1):
- Northern Illinois University, DeKalb, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw, de-identified data will be available by the researchers upon request.
Supporting Information: Study Protocol, SAP, ICF